CLINICAL TRIAL: NCT02450253
Title: Perfusion by Arterial Spin Labelling Following Single Dose Tadalafil in Small Vessel Disease (PASTIS) Trial
Acronym: PASTIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Alzheimer's Society (Other); University of Copenhagen (Other); University of Glasgow (Other); St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 14.0189; 2015-001235-20 (EudraCT Number); 15/LO/0714 (Other: Research Ethics Committee (REC)); 20140901 (Other Grant/Funding Number: ADDF)
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2018-08

CONDITIONS: Dementia, Vascular
Keywords: Vascular cognitive impairment
MeSH Terms: conditions — Dementia, Vascular | interventions — Tadalafil; Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Active Comparator): Tadalafil 20mg Capsule Stat single dose 2 x MRI scans (pre and post dose) Neuropsychological tests pre and post IMP dose Cognitive functioning prior to 1st MRI scan of that visit
  Interventions: Drug: Tadalafil; Behavioral: Cognitive functioning tests; Behavioral: Neuropsychological tests; Other: MRI Scan - Arterial Spin Labelling
- Control (Placebo Comparator): Matched placebo Capsule Stat single dose 2 x MRI scans (pre and post dose) Neuropsychological tests pre and post IMP dose Cognitive functioning prior to 1st MRI scan of that visit
  Interventions: Drug: Placebo; Behavioral: Cognitive functioning tests; Behavioral: Neuropsychological tests; Other: MRI Scan - Arterial Spin Labelling

INTERVENTIONS:
Drug: Tadalafil — single dose, 20 mg capsule p.o.
  Other Names: Cialis
  Arms: Active Treatment
Drug: Placebo — single dose, matching capsule p.o.
  Arms: Control
Behavioral: Cognitive functioning tests — Cognitive function tests will be performed prior to MRI scan 1 performed prior to IMP dosing on 2 occasions as patient will act as their own control
  Other Names: TOPF, NIHSS, MoCA,
Behavioral: Neuropsychological tests — Neuropsychological tests will be performed prior to pre IMP dose MRI scan & then parallel V2 of the tests repeated 3-5 post IMP dose and before 2nd MRI scan.
  Participants act as own controls as 1 IMP occasion will be placebo- 2nd IMP occasion will be active. 7-30 days apart
  Other Names: CANTAB, BMIPB, RBANS subtest
Other: MRI Scan - Arterial Spin Labelling — Pre and post IMP dose on 2 occasions to detect difference in blood flow in deep brain 4 MRI scans in total

SUMMARY:
Could Tadalafil improve blood flow in deep brain tissue and potentially improve cognitive function in patients with cerebral small vessel disease

DETAILED DESCRIPTION:
Cerebral small vessel disease (SVD) is the primary cause of vascular cognitive impairment (VCI), which in its most severe form manifests as vascular dementia (VaD). SVD is a fibrous thickening of small penetrating arteries in deep brain nuclei (basal ganglia, thalami) and subcortical white matter.Clinical studies suggest that pure VCI/VaD contributes approximately 8-15% of dementia in older people Reduced CBF is well established in VCI. Improved blood flow in the vasculature of the deep white and grey matter is therefore an attractive mechanism for slowing the pathology of VCI and is a valuable biomarker for an initial proof of concept study.

To increase the likelihood of success in a full scale clinical trial of tadalafil in VCI, this study will test the effects of single dose tadalafil on cerebral blood flow in subjects with SVD using ASL-MRI. A strict definition of SVD will be used that combines clinical and MRI criteria.

Phosphodiesterase-5 (PDE5) specifically degrades cGMP within cells; limiting activation of protein kinase G. Guanylyl cyclase enzymes generate cGMP, downstream from NOS-nitric oxide signalling.

PDE5 inhibitors in SVD. PDE5 blockade is a plausible strategy to improve local cerebral blood flow (CBF), in the deep brain areas afflicted by SVD. By augmenting the NO-cGMP-PKG pathway, PDE5i drugs are expected to be vaso-relaxant in small artery myocytes.

In patients with pulmonary hypertension sildenafil improved cerebral vascular reactivity in response to hypercapnic challenge, indicative of an improvement in neurovascular coupling. Similar increased reactivity was recorded 60 min after administration of sildenafil in ED patients. By contrast, healthy volunteers showed no change in MCA blood flow following sildenafil, similar to healthy rodents, where vasodilation occurred only at high concentrations of drug. Overall it appears that PDE5i may have little effect on "healthy" cerebral arteries in rodents and humans.

Prior human studies have been single dose studies of PDE5i in healthy humans, have only used sildenafil and have in general estimated CBF from Middle Cerebral Artery (MCA) blood flow using Trans Cranial Doppler (TCD). MCA blood flow may not reflect local blood flow in the microvasculature of the deep white and deep grey matter. One study examined the effect of single dose sildenafil on CBF using SPECT in patients with vascular risk factors with or without a history of stroke. Non-stroke patients exhibited an overall increase in CBF. However, no distinction was made in this study between large vessel and lacunar stroke.

In summary, pre-clinical studies support a CBF-enhancing action of PDE5i in cerebrovascular disease, while human studies to date have been limited to sildenafil and have not specifically addressed effects on CBF in people with SVD.

Tadalafil (Cialis®) is widely-used as an oral agent for sexual dysfunction. As an inhibitor of the enzyme PDE5, tadalafil has a well-established pharmacological profile as a small vessel vasodilator. Side-effect profile and pharmacokinetics are well known and the drug is well-tolerated in the target population, over a range of oral doses and regimens. The choice of tadalafil over other PDE5 inhibitors (such as sildenafil, Viagra®) is based on potency, selectivity for PDE5, plasma half-life and documented brain penetration.

Phosphodiesterase-5 (PDE5) specifically degrades cGMP within cells; limiting activation of protein kinase G. Guanylyl cyclase enzymes generate cGMP, downstream from NOS-nitric oxide signalling. The PDE5 inhibitor sildenafil (Viagra®; discovered at Pfizer, Sandwich UK) raised the profile of PDE5 as a therapeutic target. Tadalafil (Cialis®; licence holder: Eli Lilly) is widely prescribed on an "as required" basis for ED in men. It is also licensed for regular daily use at a dose of 5 mg for benign prostatic hyperplasia and 40 mg for pulmonary hypertension. Tadalafil is well tolerated and its side effect profile is well-established

ELIGIBILITY:
Inclusion Criteria:

1. Radiological evidence of cerebral small vessel disease defined as: MRI evidence of lacunar infarct(s) (≤ 1.5 cm maximum diameter) and/or confluent deep white matter leukoaraiosis (≥ grade 2 on Fazekas scale)

2. Clinical evidence of cerebral small vessel disease can be:

1. lacunar stroke syndrome with symptoms lasting >24 hours, occurring at least 6 months previously; OR:
2. transient ischaemic attack lasting < 24 hours with limb weakness, hemi-sensory loss or dysarthria at least 6 months previously AND with MRI DWI performed acutely showing lacunar infarction, OR if MRI is not performed within 10 days of TIA, a lacunar infarction in an anatomically appropriate position is demonstrated on a subsequent MRI

   3. Age ≥ 55 years.

   4. Imaging of the carotid arteries with Doppler ultrasound, CT angiography or MR angiography in the previous 12 months, demonstrating < 70% stenosis in both internal carotid arteries

   Exclusion Criteria:
   1. Known diagnosis of dementia
   2. Cortical infarction (>1.5 cm maximum diameter)
   3. Systolic BP <90 and/or diastolic BP < 50
   4. Creatinine Clearance<50ml/min
   5. Severe hepatic impairment
   6. History of Lactose intolerance
   7. Concomitant use of PDE5 inhibitors e.g. sildenafil, tadalafil, vardenafil.
   8. Concomitant use of alpha-blockers e.g. alfuzosin, doxazosin, indoramin, prazosin, tamsulosin, and terazosin can all increase the risk of postural hypotension.
   9. Participants receiving nicorandil and nitrates e.g. isosorbide mononitrate, isosorbide dinitrate, glyceryl trinitrate
   10. weight > 130kg

   11 Uncontrolled cardiac failure

   12. Persistent or paroxysmal atrial fibrillation

   13. History of gastric ulceration

   14. History of 'sick sinus syndrome' or other supraventricular cardiac conduction conditions such as sinoatrial or atrioventricular block

   15. Uncontrolled COPD

   16. Stroke or TIA within the last 6 months

   17. MRI not tolerated or contra-indicated : MRI exclusion criteria -Participant has a cardiac pacemaker; recent surgery; vascular clips; metal implants or joint replacements; have had metal fragments in their eyes; has ever worked on a lathe; has shrapnel from a war injury; possibility of pregnancy

   18. Known monogenic causes of stroke e.g.. CADASIL

   19 Unable to provide informed consent

   20. enrolled in another CTIMP study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
change in deep brain blood flow as measured by MRI-Arterial Spin Labelling | 3-5 hours following IMP dosing

SECONDARY OUTCOMES:
Change in regional CBF in cortical grey matter areas Plasma [drug concentration] dependence of deep CBF as measured by MRI ASL Changes in neuropsychological parameters including attention in Neuro attention and cognitive speed | 3-5 hours following IMP dosing

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Dr Isaacs, MRCP PhD, Principal Investigator — St George's University Hospitals NHS Foundation Trust
Locations (1):
- St George's Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Pauls MMH, Binnie LR, Benjamin P, Betteridge S, Clarke B, Dhillon MK, Ghatala R, Hainsworth FAH, Howe FA, Khan U, Kruuse C, Madigan JB, Moynihan B, Patel B, Pereira AC, Rostrup E, Shtaya ABY, Spilling CA, Trippier S, Williams R, Young R, Barrick TR, Isaacs JD, Hainsworth AH. The PASTIS trial: Testing tadalafil for possible use in vascular cognitive impairment. Alzheimers Dement. 2022 Dec;18(12):2393-2402. doi: 10.1002/alz.12559. Epub 2022 Feb 8. PMID 35135037
- [Derived] Binnie LR, Pauls MMH, Benjamin P, Dhillon MK, Betteridge S, Clarke B, Ghatala R, Hainsworth FAH, Howe FA, Khan U, Kruuse C, Madigan JB, Moynihan B, Patel B, Pereira AC, Rostrup E, Shtaya ABY, Spilling CA, Trippier S, Williams R, Isaacs JD, Barrick TR, Hainsworth AH. Test-retest reliability of arterial spin labelling for cerebral blood flow in older adults with small vessel disease. Transl Stroke Res. 2022 Aug;13(4):583-594. doi: 10.1007/s12975-021-00983-5. Epub 2022 Jan 26. PMID 35080734